CLINICAL TRIAL: NCT03196141
Title: Perioperative Clinical Utilization of Somatic Tissue Oxygen Saturation Monitoring in Pregnant Women
Brief Title: Utilization of Somatic Tissue Oxygen Saturation Monitoring in Pregnant Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not able to recruit enough participants.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000020110
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: 3 groups: healthy volunteers (15) and normotensive (10) and pre-eclamptic (10) pregnant women during their visit to labor floor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Healthy volunteers (Active Comparator): Part#1: 15 healthy volunteers; 2 assessment sessions. Session 1: StO2 vs. EndoPAT Method comparison analysis; both StO2 and EndoPAT will be applied simultaneously & pulse oximeter probes placed bilaterally on fingers. Baseline readings will be taken for 5 minutes. The blood pressure cuff will be inflated to suprasystolic pressure and StO2 and pulsatile volume changes will be measured by peripheral arterial tonometry, continuous measurement for 3 min and repeated every 10 minutes for 3 sessions.
  Session 2: This session will occur within 1 week of session 1. This session is to determine the consistency of the response.
  All probes will be applied as in session 1 and cycles of 10 minutes for 3 sessions will be done. All the measurements in session 1 will be captured in session 2.
  This will determine inter-day variability. (total time is 53 min).
  Interventions: Diagnostic Test: StO2 and EndoPAT
- Pregnant women with normal BP (Active Comparator): Part #2: 20 participants, 10 normotensive and 10 pre-eclamptic pregnant women during their visit to labor floor.
  Session 1: Both StO2 and EndoPAT will be applied simultaneously to the same arm below a BP cuff. Baseline readings will be taken for 5 minutes, the blood pressure cuff will be inflated to suprasystolic pressure StO2 and pulsatile volume changes will be measured by peripheral arterial tonometry, continuous measurement for 3 min and repeated every 10 minutes for 3 sessions.
  Additionally, vascular stiffness with be measured by SphygmoCor to measure pulse wave velocity (PWV).
  Participants must also agree to participate OB/GYN biobanking protocol HIC# 1601017004 to be in this study.
  All participants will have follow-up at 48 hours, including a blood draw, assessment of endothelial function and vascular stiffness.
  Interventions: Diagnostic Test: StO2 and EndoPAT
- Pregnant women with high BP (Active Comparator): Part #2: 20 participants, 10 normotensive and 10 pre-eclamptic pregnant women during their visit to labor floor.
  Session 1: Both StO2 and EndoPAT will be applied simultaneously to the same arm below a BP cuff. Baseline readings will be taken for 5 minutes, the blood pressure cuff will be inflated to suprasystolic pressure StO2 and pulsatile volume changes will be measured by peripheral arterial tonometry, continuous measurement for 3 min and repeated every 10 minutes for 3 sessions.
  Additionally, vascular stiffness with be measured by SphygmoCor to measure pulse wave velocity (PWV).
  Participants must also agree to participate OB/GYN biobanking protocol HIC# 1601017004 to be in this study.
  All participants will have follow-up at 48 hours, including a blood draw, assessment of endothelial function and vascular stiffness.
  Participants with hypertension will be followed in conjunction with routine clinical follow-up at 2, 6 and 12 weeks post-partum.
  Interventions: Diagnostic Test: StO2 and EndoPAT

INTERVENTIONS:
Diagnostic Test: StO2 and EndoPAT — * StO2 probe is a lightweight plastic probe that will be applied over the brachioradilalis muscle (anterolatereal aspect of the forearm) where there is less subcutaneous fat and taped in place.
  * The EndoPAT probe will be place on a finger on the same arm.
  * Pulse oximeter probes will be connected to a finger on each hand.

SUMMARY:
The purpose of this study is to compare 3 methods of assessing endothelial function in healthy female volunteers and pregnant women with and without pregnancy induced hypertension. The methods under comparison are simultaneous tissue oxygen saturation (StO2), EndoPAT and Sphygmocor (pregnant women only). 35 participants (15 healthy, 10 pregnant normal blood pressure, 10 pregnant with hypertension) will be enrolled.

DETAILED DESCRIPTION:
In both normotensive women and others with pregnancy induced hypertension, in previous research simultaneous tissue oxygen saturation (StO2) were measured in both forearms, with a blood pressure cuff above the tissue oximetry probe on one side.

StO2 values were continuously monitored on each side during unilateral blood pressure (BP) cuff inflation (to suprasystolic pressure for 3 min), and then during deflation. Despite similarity in the forearm StO2 decline observed with cuff inflation in all women, the rise following cuff deflation - indicative of reactive hyperemia - appeared reduced in hypertensive patients, suggesting a relationship with impaired endothelial reserve.

ELIGIBILITY:
Inclusion Criteria:

Non-pregnant group:

1. > 18 years of age
2. Male or female

Pregnant group:

1. > 18 years of age
2. Pregnant women > 20 weeks
3. Diagnosis of Pre-eclampsia characterized as Systolic BP > 140 mmHg, diastolic BP > 90 mmHg after 20 weeks of gestation accompanied by new onset of proteinuria.
4. Normotensive, not meeting criteria in #3

Exclusion Criteria:

Non-pregnant group:

1. Raynaud's Disease
2. Adhesive tape allergy
3. Recent Myocardial Infarction (< 3 months)
4. Congestive Heart Failure

Pregnant group:

1. Raynaud's Disease
2. Adhesive tape allergy
3. Recent Myocardial Infarction (< 3 months)
4. Congestive Heart Failure
5. Hemodynamically unstable (SBP < 90 mmHg)
6. Fetal distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
StO2 | Baseline
  Measurement of forearm StO2 during routine cycling of a blood pressure cuff can provide a continuous index of endothelial functional reserve. Baseline measures are collected in healthy and pregnant participants.
StO2 | 48 Hours (Postpartum)
  Measurement of forearm StO2 during routine cycling of a blood pressure cuff can provide a continuous index of endothelial functional reserve. This will only be measured in pregnant participants.
Endopat | Baseline
  Measurement of Endopat during routine cycling of a blood pressure cuff can provide a continuous index of endothelial functional reserve. Baseline measures are collected in healthy and pregnant participants.
Endopat | 48 Hours (Postpartum)
  Measurement of Endopat during routine cycling of a blood pressure cuff can provide a continuous index of endothelial functional reserve. This will only be measured in pregnant participants.
SphygmoCor | Baseline
  SphygmoCor is a measurement of vascular stiffness. This will only be measured in pregnant participants.
SphygmoCor | 48 Hours (Postpartum)
  SphygmoCor is a measurement of vascular stiffness. Baseline measures are collected in healthy and pregnant participants.

SECONDARY OUTCOMES:
StO2 | 2, 6, 12 weeks (Postpartum)
  Measurement of forearm StO2 during routine cycling of a blood pressure cuff can provide a continuous index of endothelial functional reserve. This will only be measured in hypertensive pregnant participants.
Endopat | 2, 6, 12 weeks (Postpartum)
  Measurement of Endopat during routine cycling of a blood pressure cuff can provide a continuous index of endothelial functional reserve. This will only be measured in hypertensive pregnant participants.
SphygmoCor | 2, 6, 12 weeks (Postpartum)
  SphygmoCor is a measurement of vascular stiffness. This will only be measured in hypertensive pregnant participants.

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Alilan, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No